CLINICAL TRIAL: NCT04965363
Title: Prevalence of Internet Addiction and Internet Gaming Disorder Among Assiut University Students
Brief Title: Prevalence of IA and IGD Disorders Among Assiut University Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Ahmed Osman, specialist of psychiatry at neurology and psychiatry department, Assiut University
Other Study IDs: IA & IGD in Assiut university
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Internet Addiction; Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional

SUMMARY:
identifying the Prevalence of internet addiction and internet gaming disorder among Assiut university students

DETAILED DESCRIPTION:
Internet activities and technologies that are increasing rapidly have attracted young adults, leading to excessive use of the Internet and maladaptive Internet attitude known as "Internet addiction". The term "addiction", even traditionally utilized to describe a physical dependence of substances, has been applied to the excessive use of the Internet . Internet addiction disorder is expressed as too much computer use that contradicts daily activities and can harm daily function .

Internet gaming disorder (IGD) was included as a nonsubstance addiction in the appendix of the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) published in 2013 by the American Psychiatric Association. The need to add IGD to this diagnostic manual was identified by an international expert working group that reviewed over 250 articles, some of which showed the detrimental effects of excessive gaming . As part of the DSM-5 approach to defining IGD, draft diagnostic criteria were proposed with some similarities to substance use disorders and added to the appendix of the DSM-5 manual, suggesting IGD was a condition warranting further research. The harmful consequences of excessive gaming were also recognized by the World Health Organization (WHO), and gaming disorder (GD) was included in their 2018 release of the 11th revision of the International Classification of Diseases (ICD-11) .

ELIGIBILITY:
Inclusion Criteria:

* Assiut university student Active Internet user since at least 1 year Willing to give consent and complete the questionnaire

Exclusion Criteria:

* Not willing to give consent and complete the questionnaire

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Assiut university students from different practical and theoretical faculties
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
identification of the Prevalence of internet addiction and internet gaming disorder among Assiut university students using Young's Internet Addiction Test (YIAT) Internet Gaming Disorder 20 test: Arabic version | baseline
  Young's Internet Addiction Test (YIAT) is a scale developed by Young which measures the presence and severity of internet dependency among adults and The IGD-20 Test was the first standardized psychometric tool to assess Internet Gaming Disorder (IGD) according to the nine Internet Gaming Disorder (IGD) criteria as suggested by the American Psychiatric Association in the latest edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5)

SECONDARY OUTCOMES:
determination of severity of internet addiction among Assiut university students | baseline
  Young's Internet Addiction Test (YIAT) is a scale developed by Young which measures the presence and severity of internet dependency among adults and classify them into none, mild, moderate and severe

REFERENCES:
- [Background] Byun S, Ruffini C, Mills JE, Douglas AC, Niang M, Stepchenkova S, Lee SK, Loutfi J, Lee JK, Atallah M, Blanton M. Internet addiction: metasynthesis of 1996-2006 quantitative research. Cyberpsychol Behav. 2009 Apr;12(2):203-7. doi: 10.1089/cpb.2008.0102. PMID 19072075
- [Background] Block JJ. Issues for DSM-V: internet addiction. Am J Psychiatry. 2008 Mar;165(3):306-7. doi: 10.1176/appi.ajp.2007.07101556. No abstract available. PMID 18316427
- [Background] Vahia VN. Diagnostic and statistical manual of mental disorders 5: A quick glance. Indian J Psychiatry. 2013 Jul;55(3):220-3. doi: 10.4103/0019-5545.117131. No abstract available. PMID 24082241
- [Background] Petry NM, Rehbein F, Gentile DA, Lemmens JS, Rumpf HJ, Mossle T, Bischof G, Tao R, Fung DS, Borges G, Auriacombe M, Gonzalez Ibanez A, Tam P, O'Brien CP. An international consensus for assessing internet gaming disorder using the new DSM-5 approach. Addiction. 2014 Sep;109(9):1399-406. doi: 10.1111/add.12457. Epub 2014 Jan 23. PMID 24456155
- [Background] Saunders JB, Hao W, Long J, King DL, Mann K, Fauth-Buhler M, Rumpf HJ, Bowden-Jones H, Rahimi-Movaghar A, Chung T, Chan E, Bahar N, Achab S, Lee HK, Potenza M, Petry N, Spritzer D, Ambekar A, Derevensky J, Griffiths MD, Pontes HM, Kuss D, Higuchi S, Mihara S, Assangangkornchai S, Sharma M, Kashef AE, Ip P, Farrell M, Scafato E, Carragher N, Poznyak V. Gaming disorder: Its delineation as an important condition for diagnosis, management, and prevention. J Behav Addict. 2017 Sep 1;6(3):271-279. doi: 10.1556/2006.6.2017.039. Epub 2017 Aug 17. PMID 28816494
- [Background] Hawi NS. Arabic validation of the Internet addiction test. Cyberpsychol Behav Soc Netw. 2013 Mar;16(3):200-4. doi: 10.1089/cyber.2012.0426. Epub 2013 Feb 26. PMID 23441685
- [Background] Pontes HM, Kiraly O, Demetrovics Z, Griffiths MD. The conceptualisation and measurement of DSM-5 Internet Gaming Disorder: the development of the IGD-20 Test. PLoS One. 2014 Oct 14;9(10):e110137. doi: 10.1371/journal.pone.0110137. eCollection 2014. PMID 25313515
- [Background] Hawi NS, Samaha M. Validation of the Arabic Version of the Internet Gaming Disorder-20 Test. Cyberpsychol Behav Soc Netw. 2017 Apr;20(4):268-272. doi: 10.1089/cyber.2016.0493. Epub 2017 Feb 21. PMID 28394210
- [Background] El-Gilany A, El-Wehady A, El-Wasify M. Updating and validation of the socioeconomic status scale for health research in Egypt. East Mediterr Health J. 2012 Sep;18(9):962-8. doi: 10.26719/2012.18.9.962. PMID 23057390
- [Background] Kessler RC, Adler L, Ames M, Demler O, Faraone S, Hiripi E, Howes MJ, Jin R, Secnik K, Spencer T, Ustun TB, Walters EE. The World Health Organization Adult ADHD Self-Report Scale (ASRS): a short screening scale for use in the general population. Psychol Med. 2005 Feb;35(2):245-56. doi: 10.1017/s0033291704002892. PMID 15841682
- See also: Addictive behaviours: Gaming disorder — https://www.who.int/news-room/q-a-detail/addictive-behaviours-gaming-disorder
- See also: internet addiction test — http://netaddiction.com/internet-addiction-test/